CLINICAL TRIAL: NCT03169855
Title: Validation of Mesopic and Photopic Contrast Vision Tests With Respect to Nighttime Driving Ability (ContrastVal) - Influence of Dynamic Glare on (Aged) Motorist (With/Without Media Opacities)
Brief Title: Validation of Mesopic and Photopic Contrast Vision Tests With Respect to Nighttime Driving Ability
Acronym: ContrastVal
Status: Completed | Type: Observational
Sponsor: Aalen University (Other)
Collaborators: DGUV (Deutsche Gesetzliche Unfallversicherung/German Social Accident Insurance Institutions) (Unknown); Study Course Ophthalmic Optics and Optometry, University of Applied Sciences Aalen (Unknown); Study Course Mechatronics, University of Applied Sciences Aalen (Unknown); Steinbeis Transferzentrum AWFE, University of Applied Sciences Aalen (Unknown); Würzburg Institute for Traffic Sciences GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: F-2015-044#A1
Record Dates: First submitted 2017-05-19; First posted 2017-05-30 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Cataract; Traffic Accident; Vision Disorders; Driving Impaired
Keywords: Traffic Ophthalmology; Glare; Cataract; Nighttime driving; contrast sensitivity; mesopic vision
MeSH Terms: conditions — Cataract; Vision Disorders | interventions — Slit Lamp Microscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Refractive media opacities: present: Refractive media opacities: present
- Refractive media opacities: absent: Refractive media opacities: absent
  Interventions: Diagnostic Test: Slit lamp (LOCS III Score)

INTERVENTIONS:
Diagnostic Test: Slit lamp (LOCS III Score) — Diagnostic procedure only
  Other Names: Oculus Pentacam (Scheimpflug procedure, densitometry)
  Groups: Refractive media opacities: absent

SUMMARY:
A) The main purposes of this study are (i) to develop a related virtual reality (VR) environment in order to judge the nighttime driving ability under mesopic and under glare conditions (ophthalmologically healthy subjects and patients with incipient to intermediate cataract, i.e. opacities of the human lens, will participate in this study), (ii) to validate the above-mentioned VR environment with respect to a related on-road driving scenario under mesopic and glare conditions, (iii) to validate clinical photopic and mesopic contrast vision tests and glare tests with respect to the prediction of nighttime driving ability, (iv) to assess the test retest reliability of clinical photopic and mesopic contrast vision tests

B) Background:

An intact mesopic vision and a glare sensitivity within a normal range are essential pre-requisites for safe driving at nighttime (DOG & BVA, 2011). Anderson & Holiday (1995) have shown that (simulated) opacities of the refractive media (with only minor effects on daytime visual acuity) induce a pronounced impairment of contrast sensitivity under nighttime conditions. Especially under glare conditions by the headlights of traffic on the opposite lane or by stationary street illumination, an impairment of the mesopic vision may cause traffic hazards. The prevalence of impairments of the central visual acuity, the mesopic vision and the glare sensitivity is significantly higher for subjects being involved in nighttime traffic accidents (Lachenmayr, 1998). Furthermore, these impairments occur more frequently in aged drivers and are, among others, related to an increase of age-related media opacities (Aulhorn & Harms, 1970, Babizhayev, 2003). Due to the demographic change, the relevance of nighttime driving ability is increasing in the next years since more and more aged employees will participate at the motorized traffic at night.

The German Fahrerlaubnisverordnung (FEV i.e. driving license regulation) specifies pass/fail criteria with regard to mesopic vision and glare sensitivity. The luminance level during nighttime driving is usually between 0.01 and 1 cd/m^2, and therefore can be attributed to the level of mesopic vision. However, over the last years, the attempt was made to introduce photopic contrast sensitivity test to diagnose nighttime driving ability (i.e. testing of contrast vision under daytime conditions without time consuming adaptation procedures). Current research aims at investigating the relationship between contrast tests under various luminance conditions (Wilhelm et al, 2013). It is questionable, whether photopic tests are at all reliable predictors with regard to nighttime driving (Gramberg-Danielsen et al., 1984, Hertenstein et al., Graefe´s Archive of Ophthalmology, 2016).

DETAILED DESCRIPTION:
Subjects and Methods Adult patients with a distant binocular visual acuity of ≥ 0.8 (≥ 16/20; habitual correction) and healthy control subjects will be included in this explorative study after informed consent.

The study will be subdivided in the following (three) parts:

Part 1: Validation of the Aalen driving simulator set-up (ten patients with incipient to moderate cataract, i.e. opacities of the human lens of varying localization and of various degree of expression in at least one eye and ten age- and gender-correlated ophthalmologically healthy control subjects will be enrolled) Part 1.1.: Comprehensive ophthalmological/optical examination (Aalen University of Applied Sciences) including a detailed ophthalmological and medical history.

Part 1.2.: Baseline driving simulator test under mesopic conditions with/without glare under simulated static/simulated driving conditions (Aalen University of Applied Sciences) Part 1.3.: Baseline on road test under mesopic conditions with/without glare, under on road static/on road driving conditions (Aalen University of Applied Sciences) (If possible, the sequence of Part 1.2. and Part 1.3. will be randomly assigned.)

Part 2: Advanced driving simulator test (twenty patients with incipient to moderate cataract, i.e. opacities of the human lens of varying localization and of various degree of expression in at least one eye and twenty age- and gender-correlated ophthalmologically healthy control subjects will be enrolled. Subjects being enrolled in Part 1, will be asked to participate also at Part 2 and Part 3.) Part 2.1.: Comprehensive ophthalmological/optical examination of all (newly) enrolled patients and subjects who have not already been examined in Part. 1.1. (Aalen University of Applied Sciences).

Part 2.2.: Advanced driving simulator test under photopic and under mesopic simulated driving with and without glare (Würzburg Institute for Traffic Sciences = WIVW) in order to investigate the influence of glare on the driving behavior

Part 3: Representative driving simulator test (The [altogether fourty] subjects, enrolled in Part 2, will be enrolled in this part of the study.) Driving simulator test under photopic and mesopic conditions in oder to investigate glare on representative driving situations. Driving performance will be evaluated highly-standardized and partially automated on different parameters of operational and tactical driving behavior (S.A.F.E., Würzburg Institute for Traffic Sciences = WIVW).

Pass/fail rates are specified as described in the related manuals of the instruments. With regard to visual acuity measurements and assessment of mesopic contrast vision without/with glare, results are rated according to DIN 58220 - Part 3/ISO 10938: If less than three out of five subsequent presentations of an eight-position LANDOLT C (with two oblique and three horizontal/vertical gap locations in random sequence) are correctly identified, the session is rated as failed. Overlooking/missing reactions to obstacles (pedestrian [display dummy with dark clothing]/wild boar at the right roadside) are rated as failed.

For mesopic contrast vision testing, single LANDOLT optotpyes (visual acuity level 0.1 = 2/20) with the contrast levels (1:2, 1:5 and 1:23, respectively, according to AULHORN/HARMS) are presented via the Optovist Instrument (Vistec, Inc., Manching/Germany) or via the head up display (HUD) of the simulator vehicle/on road vehicle.

Photopic and mesopic contrast vision tests (without glare) are repeated once in order to assess the test retest variability of the related test procedure.

1. LANDOLT C chart for presentation of high contrast optotypes according to DIN 58220 - Part 3/ISO 10938 (Visus GmbH, Stuttgart/Germany)
2. Assessment of low contrast visual acuity using FrACT (Freiburg Visual Acuity Test, internet version 3.8.1)
3. Assessment of photopic contrast sensitivity, using the MARS Letter Contrast Sensitivity Test (The Mars Perceptrix Corporation, NY 10514-2523,USA)
4. Assessment of mesopic contrast sensitivity, using the OPTOVIST (VISTEC, Manching/FRG)
5. Judgment of intraocular straylight, using the C-Quant (Straylight meter, OCULUS, Dutenhofen/FRG)
6. Classification of human crystalline lens opacities, using the BQ 900 slitlamp (HAAG-STREIT, Köniz/CH), digital photography with dilated pupils, applying the LOCS III score
7. Densitometry of the crystalline lens, using the Pentacam HR (OCULUS Inc., Dutenhofen/FRG)
8. Digital Fundus Photography with dilated pupils (WX3D fundus camera, KOWA Optimed Deutschland GmbH, Düsseldorf/FRG)
9. Aalen driving simulator: Two high performance VELVET planetarium projectors (Fa. ZEISS, Jena/FRG), AUDI A4 (AUDI Inc., Ingolstadt/FRG) with digital display and re-equipped (BFFT, Gaimersheim/FRG) with externally controllable head up display (HUD) for presentation of LANDOLT Cs with varying contrast levels, SILAB virtual reality environment (WIVW, Veitshöchheim/FRG), two mobile glare sources (LED arrays)
10. Aalen on road parcours: AUDI A4 (AUDI Inc., Ingolstadt/FRG) with digital display, with externally controllable head up display (HUD, VW AG, Wolfsburg/FRG)) for presentation of LANDOLT Cs with varying contrast levels and equipped with dual brake (VEIGEL GmbH + Co KG, Künzelsau/FRG)

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years (preferred: age, exceeding 50 yrs.)
* Minimum distant visual acuity (with habitual correction) 0.8 (16/20, single optotypes, LANDOLT C chart for presentation of high contrast optotypes according to DIN 58220 - Part 3/ISO 10938 (Visus GmbH, Stuttgart/Germany)
* ametropia maximum spherical ametropia sph ±8.00 dpt maximum maximum astigmatism cyl 2.00 dpt
* normal (age-corrected) visual field
* clear refractive media OR incipient to intermediate cataract
* informed consent

Exclusion Criteria:

* epilepsy / psychiatric disorders
* drugs, interfering with reaction time and/or with visual acuity or with refractive status of the eye
* deficient driving license
* yearly mileage less than 3000 km/y (less than 1.864 miles/y)

ophthalmological exclusion criteria: all ophthalmological diseases or abnormalities, with the exception of those, listed in the above-mentioned inclusion criteria

* amblyopia
* strabismus
* ocular motility disorders
* nystagmus
* double vision
* albinism
* glaucoma / IOP exceeding 22 mmHg
* shallow anterior chamber/risk of angle closure glaucoma (van HERICK grade less than 2)
* macular diseases / maculopathy
* diabetic retinopathy (blood sugar-related retinal disease)
* status post severe eye injuries
* eye surgery within the last three months (, related to the time point of recruitment)
* Infectious diseases (conjunctivitis, corneal inflammation, uveitis)
* very dry eyes (sicca symptoms)
* drugs inducing miosis
* any other eye disorders that affect the image quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ophthalmologically healthy subjects and patients with incipient to intermediate cataract.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Pass/fail rate (i.e. ratio of "no. of subjects passed" by "total no. of participants") with respect to a vision-related driving ability test | From date of "first subject in" to date of "last subject out", i.e. over an 18 months period
  Pass/fail rates will be assessed for vision related driving ability tests:
  (i) clinical photopic/mesopic contrast vision tests, (ii) glare tests, (iii) of driving simulator tests under mesopic conditions with and without glare, and (iv) on-road tests under mesopic conditions with and without glare

SECONDARY OUTCOMES:
Rank of tested subjects with respect to a vision-related driving ability test | From date of "first subject in" to date of "last subject out", i.e. over an 18 months period
  Rank/i.e. sequence of tested subjects with respect to the results of a vision-related driving ability test [see clauses (i) to (iv), Outcome 1]
Test-retest reliability, expressed as "limits of agreement" (LOA) of a clinical contrast vision test | From date of "first subject in" to date of "last subject out", i.e. over an 18 months period
  Test-retest reliability of a clinical photopic/mesopic contrast vision test [see clauses (i) and (ii), Outcome 1]
Response time (in milliseconds) regarding to the gap recognition of a standardized optotype | From date of "first subject in" to date of "last subject out", i.e. over an 18 months period
  Response time regarding gap recognition of a standardized optotype (8 position LANDOLT C) with three contrast levels, presented via the head up display
Intensity of driving simulator sickness, assessed by a questionnaire | From date of "first subject in" to date of "last subject out", i.e. over an 18 months period
  Intensity of driving simulator sickness, assessed by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schiefer, Prof. Dr., Principal Investigator — Aalen University of Applied Sciences
Locations (1):
- University of Applied Sciences, Study Course Ophthalmic Optics, Aalen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No